CLINICAL TRIAL: NCT01290042
Title: A Phase 1, Randomized, Double-Blind, Placebo-controlled, Ascending Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 181 in Healthy Subjects, in Subjects With Active Ulcerative Colitis, and in Subjects With Active Crohn's Disease.
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 181.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20101261
Record Dates: First submitted 2011-01-27; First posted 2011-02-04 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — abrilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo arm (Active Comparator): Four escalating dose levels of AMG 181 administered as multiple doses of AMG 181 in healthy subjects, in subjects with active ulcerative colitis, and in subjects with active Crohn's disease.
  Interventions: Other: Placebo for AMG 181
- Active arm (Active Comparator): Four escalating dose levels of AMG 181 administered as multiple doses of AMG 181 in healthy subjects, in subjects with active ulcerative colitis, and in subjects with active Crohn's disease.
  Interventions: Drug: AMG 181

INTERVENTIONS:
Drug: AMG 181 — Four escalating dose levels of AMG 181 administered as multiple doses of AMG 181 in healthy subjects, in subjects with active ulcerative colitis, and in subjects with active Crohn's disease.
  Arms: Active arm
Other: Placebo for AMG 181 — Four escalating dose levels of AMG 181 administered as multiple doses of AMG 181 in healthy subjects, in subjects with active ulcerative colitis, and in subjects with active Crohn's disease.
  Arms: Placebo arm

SUMMARY:
To assess the safety and tolerability of multiple subcutaneous doses of AMG 181 in healthy subjects, in subjects with active ulcerative colitis, and in subjects with active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 34 kg/m2
* Normal physical and neurological examination, clinical laboratory values and ECG
* Ulcerative Colitis Disease Activity Index (UCDAI, aka Mayo score) score of 4 to 10 (inclusive), with a minimum sigmoidoscopy score of 1; (for subjects with ulcerative colitis)
* Crohn's Disease Activity Index (CDAI) score of >150 and < 450 at screening (for subjects with Crohn's disease)
* Additional inclusion criteria apply

Exclusion Criteria:

* History or evidence of a clinically significant disorder (including psychiatric), condition or disease that would pose a risk to subject safety or interfere with the study evaluations, procedures or completion
* History of malignancy of any type, other than in situ cervical cancer or surgically excised non-melanomatous skin cancers within the past 5 years
* Underlying condition(s) that predisposes the subject to infections
* Disease limited to the rectum, i.e. within 10 cm of the anal verge (for subjects with ulcerative colitis)
* Evidence of severe disease (as evidenced by an Hb concentration less or equal to 10g/dL; toxic megacolon, or an UCDAI score greater than 10) (for subjects with ulcerative colitis)
* Subject has short bowel syndrome (for subjects with Crohn's disease)
* Presence of an ostomy (for subjects with Crohn's disease)
* Presence of a fistula (for subjects with Crohn's disease)
* Additional exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To assess the number of adverse events per subject, after multiple subcutaneous doses of AMG 181 in in healthy subjects, in subjects with active ulcerative colitis, and in subjects with active Crohn's disease. | 40 Weeks

SECONDARY OUTCOMES:
To measure the area under the plasma concentration curve versus time of drug AMG 181. | 29 Weeks
To assess receptor saturation percentages relative to baseline after multiple doses of AMG 181. | 29 Weeks
To evaluate changes in peripheral blood T lymphocyte subsets counts relative to baseline after multiple doses of AMG 181. | 29 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (5):
  - Research Site, Glendale, California
  - Research Site, Bridgeport, Connecticut
  - Research Site, Danbury, Connecticut
  - Research Site, Miami, Florida
  - Research Site, Duncansville, Pennsylvania
- Australia (3):
  - Research Site, Herston, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Prahran, Victoria

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com